CLINICAL TRIAL: NCT01572753
Title: A Single Centre, Multiple Dose, Open Label Randomised Trial to Evaluate the Effect of Post Dose Meal Timings and the Effect of Volume of Water With Dosing on the Pharmacokinetic Properties of Oral Semaglutide in Healthy Male Subjects
Brief Title: Investigation of Optimal Dosing Conditions for a Long Acting GLP-1 Analogue in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-3794; 2010-019653-17 (EudraCT Number); U1111-1120-6776 (Other: WHO)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Post-dose fasting 120 mins/50 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 60 mins/50 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 30 mins/50 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 15 mins/50 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 120 mins/120 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 60 mins/120 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 30 mins/120 ml water (Experimental)
  Interventions: Drug: semaglutide
- Post-dose fasting 15 mins/120 ml water (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 50 ml of water. During the post-dose fasting period of 120 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 120 mins/50 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 50 ml of water. During the post-dose fasting period of 60 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 60 mins/50 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 50 ml of water. During the post-dose fasting period of 30 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 30 mins/50 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 50 ml of water. During the post-dose fasting period of 15 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 15 mins/50 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 120 ml of water. During the post-dose fasting period of 120 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 120 mins/120 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 120 ml of water. During the post-dose fasting period of 60 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 60 mins/120 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 120 ml of water. During the post-dose fasting period of 30 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 30 mins/120 ml water
Drug: semaglutide — Subjects will be dosed in the morning, for 10 days, after an overnight fast (liquid will not be allowed from 2 hours before dosing). Dose to be taken with 120 ml of water. During the post-dose fasting period of 15 mins, no food or liquid is allowed.
  Arms: Post-dose fasting 15 mins/120 ml water

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to evaluate the optimal dosing conditions for semaglutide (a long acting GLP-1 analogue) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the investigator, based on medical history, physical examination, electrocardiogram (ECG), vital signs and clinical laboratory
* Body mass index (BMI) of 18.5-30.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Males who are sexually active and not surgically sterilised, who or whose partner(s): a. are not using adequate contraceptive methods (e.g. condom with spermicidal foam/gel/film/cream or contraceptives with a Pearl Index below 1%, such as implants, injectables, combined oral contraceptives, or hormonal intrauterine devices or diaphragm + spermicide) or b. do not refrain from sexual intercourse during the trial and until 30 days following the last dose of trial medication. In addition, subjects must not donate sperm for the duration of the trial and for 30 days following the last dose of trial medication or c. sterilization of either partner
* Suffer from a life threatening disease or has a history of any clinically significant disease or disorder
* History of acute idiopathic or chronic pancreatitis
* Calcitonin value equal to or above 50 ng/L
* Any clinically significant abnormal laboratory test results (haematology, biochemistry and urinalysis), as judged by the investigator and any of the following laboratory safety results (based on screening results): Amylase, lipase and creatinine, above upper normal range. Aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT) and gamma-glutamyl-transpeptidase (gamma-GT) above 1.5 times upper normal range (UNR). Thrombocytes below 0.75 times lower normal range (LNR) or above 1.25 times UNR. Leucocytes outside 3.0 to 11.0x10^9/L (normal range is 3.91 to 8.77x10^9/L. Sodium outside the range 130.0 to 150.0 mmol/L (normal range is 136-145 mmol/L). Potassium outside the range 3.0 to 5.5 mmol/L (normal range is 3.5 to 5.1 mmol/L)
* Any clinically significant abnormal ECG, as judged by the investigator
* Subjects who are smokers

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2012-09-08 (Actual); Study Completion 2012-09-08 (Actual)

PRIMARY OUTCOMES:
AUC 0-24h; Area under the semaglutide concentration curve from time 0-24 hours after the 10th dosing | 0-24hrs after the 10th dosing

SECONDARY OUTCOMES:
Cmax; The maximum plasma semaglutide concentration | Post-dose at day 10
tmax; Time to maximum plasma semaglutide concentration | Post-dose at day 10
t1/2; the terminal half-life of semaglutide | Post-dose at day 10

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Baekdal TA, Breitschaft A, Donsmark M, Maarbjerg SJ, Sondergaard FL, Borregaard J. Effect of Various Dosing Conditions on the Pharmacokinetics of Oral Semaglutide, a Human Glucagon-Like Peptide-1 Analogue in a Tablet Formulation. Diabetes Ther. 2021 Jul;12(7):1915-1927. doi: 10.1007/s13300-021-01078-y. Epub 2021 Jun 2. PMID 34080123
- [Derived] Overgaard RV, Navarria A, Ingwersen SH, Baekdal TA, Kildemoes RJ. Clinical Pharmacokinetics of Oral Semaglutide: Analyses of Data from Clinical Pharmacology Trials. Clin Pharmacokinet. 2021 Oct;60(10):1335-1348. doi: 10.1007/s40262-021-01025-x. Epub 2021 May 10. PMID 33969456
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com